CLINICAL TRIAL: NCT02455960
Title: Protective Effects of Oral L-Arginine Supplement in Patients With CKD After Intravenous Contrast Media Injection
Brief Title: Protective Effects of Oral L-Arginine CI-AKI
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Phramongkutklao College of Medicine and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Arginine 01
Record Dates: First submitted 2015-05-25; First posted 2015-05-28 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Contrast Induced AKI
MeSH Terms: interventions — Arginine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arginine (Experimental): Participants need to take arginine 3 g/day orally for 3 days before CT with contrast media injection
  Interventions: Dietary Supplement: L-arginine
- Placebo (Placebo Comparator): Participants need to take placebo (corn powder) 3 g/day orally for 3 days before CT with contrast media injection
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: L-arginine — Comparison of the efficacy of L-arginine 3 grams for days versus placebo in contrast induced AKI prevention
  Arms: Arginine
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
This trial was performed to examine the efficacy of oral L-arginine for preventing CI-AKI in chronic kidney disease (CKD) patients.

DETAILED DESCRIPTION:
Contrast-induced acute kidney injury (CI-AKI) is a common complication in hospitalized patients. Nitric oxide-signal transduction plays an important role in prevention of CI-AKI. L-Arginine is an amino acid involved in ammonia detoxification, and is well known as a precursor to nitric oxide, a key component of endothelial-derived relaxing factor.

This is a prospective randomized, double blind, placebo controlled trial among CKD stage 3-4 patients undergoing computer tomography. Eligible patients were randomly assigned to two groups: (1) arginine 3 g/day or 6 capsules per day, and (2) placebo 6 capsules per day for 3 days before contrast media injection. Serum cystatin C, serum creatinine and estimated GFR was measured at baseline and 48 hours after procedure.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Stable CKD stage 3-4 patients
* Patients undergoing elective contrast media injection

Exclusion Criteria:

* History of arginine allergy
* Acute kidney injury diagnosed within 4 weeks
* Active infection/sepsis
* Severe liver disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2014-09; Primary Completion 2016-04 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of Contrast-induced acute kidney injury (CI-AKI) | 48 hours

SECONDARY OUTCOMES:
Number of Adverse effects | 48 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Nephrology, Phramongkutklao Hospital, Rachatevee, Bangkok, Thailand